CLINICAL TRIAL: NCT06477874
Title: ASSESSMENT OF DENTAL IMPLANTS PLACED IN MANDIBULAR CONSOLIDATED ILIAC-CREST BONE GRAFTS USING DENSAH BURS VERSUS THE STANDARD DRILLS (A Randomized Controlled Trial)
Brief Title: Assessment of Implants Placed in Consolidated Graft With Different Bone Drills.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Amr Gibaly, Associate Professor of Oral and Maxillofacial Surgery, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Implant Complication; Bone Graft; Mechanical Complications
Keywords: Bone graft; Iliac crest; Implant stability

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Active Comparator): The dental implants placed after bone osseodensification using densah burs
  Interventions: Procedure: Dental implants placement
- Control group (Active Comparator): The dental implants placed after conventional bone drilling with the standard drills
  Interventions: Procedure: Dental implants placement

INTERVENTIONS:
Procedure: Dental implants placement — implants placed in consolidated bone grafts

SUMMARY:
The anterior iliac crest is a popular source of bone harvest. However, when fused to the intramembranous jaw bones, it yields low-density bones that qualitatively and quantitatively endanger the fixture's stability.

In 1994, Summers first documented using the bone-condensing approach to improve the primary stability of dental implants.

This study aims to determine whether osseodensifying the consolidated mandibular bone grafts will improve implant stability and marginal bone loss

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes with an age range of 18-55 years.
2. Patients subjected to a successful iliac crest mandibular bone graft after segmental mandibular resection.
3. A minimal ridge height of ten millimeters and a ridge width of seven millimeters.
4. Healthy soft tissue coverage, with a reasonable interaction space.

Exclusion Criteria:

1. Clinical or radiographic signs of graft infection, rejection, or massive resorption.
2. The previous exposure to radiotherapy or chemotherapy.
3. Any systemic disease that would affect bone healing or implant osseointegration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-06-09 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic bone loss | 6 months osseointegration period
  Calibration of the amplitude of vertical bone loss

SECONDARY OUTCOMES:
Implant stability | 6 months osseointegration period
  Calibration of primary and secondary implant stability quotient

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial Surgery, Faculty of Oral and Dental Medicine, Modern University for Technology & Information., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No